CLINICAL TRIAL: NCT03780647
Title: Assessment of the Impact of Thoracic Outlet Syndromes on the Performance at Work
Acronym: PROCTB
Status: Terminated | Type: Observational
Why Stopped: due to Covid19 pandemic , the inclusions slow down , and the rate of occupational problems exceeding by more than 300% changing the objective and the size of the study
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_26; 2018-A00289-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Thoracic outlet syndrome; Performance at work
MeSH Terms: conditions — Thoracic Outlet Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspicion of thoracic outlet syndrome
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Assessment of the impairment at work by a specific auto- questionnaire given after echo-Doppler that confirm the diagnosis

SUMMARY:
Thoracic outlet syndrome may associate neurologic, arterial and venous symptoms. The responsibility of repetitive movements and postural factors has been mentioned for long. Some tasks are hard to perform, and it seemed interesting to assess the consequences of this syndrome on the work capacity by a questionnaire, at the moment of diagnosis by Echo-Doppler

ELIGIBILITY:
Inclusion Criteria:

* A stenosis of at least 80% of arterial stenosis at Echo-Doppler examination during abduction-retropulsion of the arm
* Actually employed or having been employed

Exclusion Criteria:

* Cognitive or mental impairment
* Illiteracy
* Visual impairment
* Patients having been diagnosed with fibromyalgia, chronic fatigue syndrome or ehler-Danlos syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients sent to the University Hospital radiology department or to an angiologist with private practice for a suspicion of thoracic outlet syndrome, with diagnosis confirmed by Echo-Doppler
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Frequency of an impairment at work | Baseline: one session

SECONDARY OUTCOMES:
Frequency of job loss | Baseline: one session
Frequency of income loss | Baseline: one session

CONTACTS AND LOCATIONS:
Overall Officials: André THEVENON, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swynghedau, CHU, Lille, France

REFERENCES:
- [Derived] Logiou C, Demondion X, Tiffreau V, Wieczorek V, Thevenon A. Evaluation of the socioprofessional consequences of thoracic outlet syndrome. BMC Res Notes. 2023 Sep 11;16(1):207. doi: 10.1186/s13104-023-06448-2. PMID 37697402